CLINICAL TRIAL: NCT05741333
Title: Pivotal In-Office Clinical Study of the Solo+ Tympanostomy Tube Device
Brief Title: In-Office Clinical Study of the Solo+ TTD
Acronym: VENTY
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: AventaMed DAC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSP003
Record Dates: First submitted 2023-02-14; First posted 2023-02-23 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Ear Infection; Otitis Media
MeSH Terms: conditions — Otitis; Otitis Media

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Solo+ Tympanostomy Tube Device (Solo+ TTD) (Experimental): The Solo+ TTD is a disposable surgical tool designed to deliver a tympanostomy tube into the tympanic membrane of patients undergoing a tympanostomy tube placement procedure.
  Interventions: Device: Solo+ Tympanostomy Tube Device (Solo+ TTD)

INTERVENTIONS:
Device: Solo+ Tympanostomy Tube Device (Solo+ TTD) — The Solo+ TTD is intended to deliver a tympanostomy tube through the tympanic membrane of a patient.

SUMMARY:
The objective of this study is to evaluate the safety and effectiveness of the Solo+ Tympanostomy Tube Device (Solo+ TTD) for the placement of tympanostomy tubes in paediatric patients undergoing a tympanostomy procedure.

DETAILED DESCRIPTION:
The study will be a multi-site, prospective, treatment-only study to gather safety and effectiveness data on the use of the Solo+ TTD in-office with topical anesthesia in children aged ≥6 months to <13 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥6 months to <13 years
* Planned tympanostomy tube insertion
* Patient is able to commit to the follow-up visits and assessments

Exclusion Criteria:

* Anatomy that precludes sufficient visualization of the tympanic membrane
* Anatomy that precludes safe access to the tympanic membrane and safe use of the Solo+ TTD
* Narrow ear canals
* Congenital or craniofacial abnormalities affecting the ear
* No baseline audiometry or tympanometry
* Familial history of insensitivity to anesthetic components
* Patient unable to remain still or is unsuitable for protective stabilization to undergo an in-office procedure

Ages: 6 Months to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 66 (Estimated)
Dates: Start 2023-03-30 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Procedure Success | Intra-operative
  Percentage of subjects in which the Solo+ TTD tympanostomy tube is inserted in all indicated ears
Rate of Adverse Events | 24 months
  Incidence and nature of device- or procedure-related adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Matija Daniel, Study Chair — Queen's Medical Center
Locations (7):
- United States (7):
  - Southern Head & Neck Surgery, Alexander City, Alabama
  - North Alabama ENT, Huntsville, Alabama
  - East Alabama ENT, Opelika, Alabama
  - Sacramento ENT, Sacramento, California
  - Advanced ENT & Allergy, Louisville, Kentucky
  - Specialty Physician Associates, Bethlehem, Pennsylvania
  - South Carolina ENT, Columbia, South Carolina

IPD SHARING:
Plan to Share IPD: No